CLINICAL TRIAL: NCT00434473
Title: IMPACTS Trial: Investigation of the Modulation of Phospholipase in Acute Chest Syndrome (Dose Escalation Study: Varespladib Infusion [A-001] for the Prevention of Acute Chest Syndrome in At-Risk Patients With Sickle Cell Disease and Vaso-occlusive Crisis)
Brief Title: IMPACTS Trial: Investigation of the Modulation of Phospholipase in Acute Chest Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AN-SCD1121
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis; Acute Chest Syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Chest Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- A-001 (Experimental)
  Interventions: Drug: A-001

INTERVENTIONS:
Drug: A-001 — A-001
  Arms: A-001
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study will be conducted at 15-20 US centers in a randomized, placebo-controlled, double-blind fashion. Enrollees will be hospitalized sickle cell disease (SCD) patients at-risk for acute chest syndrome (ACS) based on the presence of vaso-occlusive crisis (VOC), fever (T ≥38.0°C) and serum sPLA2 concentration ≥50 ng/mL.

DETAILED DESCRIPTION:
This is a double-blind randomized, parallel group, placebo-controlled dose escalation study (2 cohorts) in patients with sickle cell disease (SCD) and vaso-occlusive crisis (VOC) who are at-risk for development of acute chest syndrome (ACS) based on the combination of VOC, fever (T ≥38.0ºC), and a serum sPLA2 concentration ≥50 ng/mL.

The first group of patients will be randomized 2:1 to receive low dose A-001 or placebo as a 48-hour continuous infusion. Pharmacokinetic and clinical data from this group will undergo review by the Independent Data Monitoring Committee (IDMC). If there is no significant toxicity associated with A-001, then an additional group of patients will be enrolled and randomized 2:1 to high dose A-001 versus placebo as a 48-hour continuous infusion.

ELIGIBILITY:
Patients are eligible for inclusion if they meet the following criteria:

* Sickle cell variant (Hb SS, Hb SC, sickle β°-thalassemia, sickle β+-thalassemia)
* Pain consistent with vaso-occlusive crisis
* Elevated serum sPLA2 level (measured on-site)
* Fever
* Age ≥5 years (through adult)

Patients must NOT meet any of the following exclusion criteria:

* New lung infiltrate by chest radiography
* Pregnancy or breastfeeding
* Significant renal dysfunction
* Significant hepatic dysfunction
* Acute neurologic dysfunction
* Any medical condition for which transfusion may be needed imminently, and/or hemoglobin <5 g/dL
* Red blood cell transfusion within 30 days of entry into the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of different doses of A 001 therapy when administered as a 2-day continuous infusion to sickle cell disease (SCD) patients at-risk for the acute chest syndrome (ACS). | Study end

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of A-001 in SCD patients | Study end
To confirm the ability of A-001 infusion to suppress serum sPLA2 activity in SCD patients with elevated serum sPLA2 | Study end
To determine the efficacy of A-001 infusion in preventing ACS in SCD patients with the combination of vaso-occlusive crisis (VOC), fever, and elevated serum sPLA2 | Study end

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Duke University Comprehensive Sickle Cell Center, Durham, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia